CLINICAL TRIAL: NCT01127074
Title: Phase 1 Study: Induction of Systemic Immune Responses in Metastatic Breast Cancer Patients by Vaccination With a CD80-modified, Devitalized HLA-*A0201+ Breast Cancer Cell Line (KS24.22)
Brief Title: Vaccination of Metastatic Breast Cancer Patients With a CD80-modified Allogeneic Cancer Cell Line (KS2422)
Acronym: KS2422-vacc
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Paul Ehrlich Institute, Langen, Germany (Unknown)
Responsible Party: Prof. D. Wallwiener, University of Tuebingen, Dep. of Obst. and Gynecology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01 KV 9540
Record Dates: First submitted 2010-05-18; First posted 2010-05-20 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2010-05

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer; breast cancer stage IV; vaccination; CD80; immunotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KS24.22-vaccination (Experimental): The first four vaccinations, which were given every two weeks, were followed by four monthly vaccinations. Additional vaccinations were permitted on request for patients who exhibited stable disease (SD).
  Immediately before administration, KS24.22 cells were thawed and lethally irradiated. KS24.22 cells were adjusted to 10E7/ml in Ringer-Lactate-solution, transferred to 1 ml syringes and stored on ice until injected within a time frame of 2h. Vaccinations were given i.d. in the thigh with a total volume of 1 ml divided between two injection sites.
  Interventions: Biological: KS24.22 cells

INTERVENTIONS:
Biological: KS24.22 cells — The first four vaccinations, which were given every two weeks, were followed by four monthly vaccinations. Additional vaccinations were permitted on request for patients who exhibited stable disease (SD).
  Immediately before administration, KS24.22 cells were thawed and lethally irradiated (200 gray). KS24.22 cells were adjusted to 107/ml in Ringer-Lactate-solution, transferred to 1 ml syringes and stored on ice until injected within a time frame of 2h. Vaccinations were given i.d. in the thigh with a total volume of 1 ml divided between two injection sites.

SUMMARY:
In the last few years there has been a great attempt to develop active immunotherapies for breast cancer patients (BCPs) using undefined as well as selected antigens to activate tumor specific T-lymphocytes. The purpose of this phase-I study was to determine the safety and feasibility of vaccinations with an allogeneic breast cancer cell line, KS24.22, genetically modified to express CD80 and Her-2/neu, and to evaluate the efficacy of inducing tumor antigen-specific immune responses in human leukocyte antigen(HLA)-A*02-matched patients with metastatic breast cancer.

DETAILED DESCRIPTION:
The trial was designed as an open label phase-I. Informed consent was given twice by the patients (1st for HLA-typing, 2nd for participation in the vaccination trial).

The first four vaccinations, which were given every two weeks, were followed by four monthly vaccinations. Additional vaccinations were permitted on request for patients who exhibited stable disease (SD).

Immediately before administration, KS24.22 cells were thawed and lethally irradiated. KS24.22 cells were adjusted to 10E7/ml in Ringer-Lactate-solution, transferred to 1 ml syringes and stored on ice until injected within a time frame of 2h. Vaccinations were given i.d. in the thigh with a total volume of 1 ml divided between two injection sites.

ELIGIBILITY:
Inclusion Criteria:

* proven diagnosis of carcinoma of the breast with distant metastatic disease
* patient received either anthracycline- or taxane-based chemotherapy ("state of the art")
* Karnofsky Score (performance status) 80%
* HLA-*A0201-positive
* minimum life expectancy of 6 month
* written informed consent
* activation of patient's T-lymphocytes by mitogen antibodies and the cell line used for vaccination

Exclusion Criteria:

* manifestation of CNS metastases
* immunosuppressive disease like AIDS, autoimmune disease
* no serious concomitant systemic medical disorders or active acute or systemic infection
* pregnancy
* chemotherapies or radiotherapies in the 4 weeks preceding study entry
* biological response modifiers (antibodies, TNF, cytokines) or other immune therapies in the 6 weeks preceding study entry (exclusion: hematopoetic growth factors)
* organ transplanted patients

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2002-03; Primary Completion 2008-07 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
safety of KS24.22 administration | 2 years
feasibility

SECONDARY OUTCOMES:
immunological response | 2 years
progression free survival
overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Diethelm Wallwiener, Principal Investigator — University Hospital Tuebingen
Locations (1):
- Univ. of Tuebingen, Dep. Obst. and Gynecology, Tübingen, Germany

REFERENCES:
- [Result] Guckel B, Stumm S, Rentzsch C, Marme A, Mannhardt G, Wallwiener D. A CD80-transfected human breast cancer cell variant induces HER-2/neu-specific T cells in HLA-A*02-matched situations in vitro as well as in vivo. Cancer Immunol Immunother. 2005 Feb;54(2):129-40. doi: 10.1007/s00262-004-0583-z. Epub 2004 Sep 9. PMID 15365776